CLINICAL TRIAL: NCT06221228
Title: Flipped Classroom Approach in Continuous Ambulatory Peritoneal Dialysis Training: Protocol
Brief Title: Flipped Classroom Approach in Continuous Ambulatory Peritoneal Dialysis Training
Acronym: FCCAPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HSEARS20230905003
Record Dates: First submitted 2023-12-20; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-11

CONDITIONS: Chronic Kidney Disease
Keywords: Continuous Ambulatory Peritoneal Dialysis Training; Pre-dialysis education programme; flipped class pedagoggy
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Training (CT): (No Intervention): Usual care in the clinical practice: Pre-dialysis training class
- Audio-visual assisted Flipped Classroom pre-dialysis training (Experimental): The audio-visual assisted Flipped Classroom (FC) CAPD Training Programme is a one-week individual intervention, which consists of five sessions (8-hours each). Pre-class audio-visual tutorials will be provided for self-study prior to F2F sessions. Six instructional videos, each dedicated to a specific procedure, are accessible for preview and repeated viewing as needed. Such flexibility allows the patients to revise at their own preferred time and pace. The four videos are (1) CAPD preparation and hand washing, (2) CAPD bag exchange procedure (Ultrabag or Balance systems), (3) Trouble shooting, and (4) Addressing contamination, (5) Detecting peritonitis, and (6) Exit site care. Participants will be asked to take note of any issues or difficulties they encounter while watching the video. A CAPD education booklet will be prepared and distributed to the patients at the beginning of the F2F training session. Take-home exercises will allow participants to revise the materials covered.
  Interventions: Behavioral: Audio-visual assisted Flipped Classroom (FC) CAPD Training Programme

INTERVENTIONS:
Behavioral: Audio-visual assisted Flipped Classroom (FC) CAPD Training Programme — FC CAPD programme is a one-week individual intervention, which consists of five sessions (8-hours each).
  Pre-class audio-visual tutorials will be provided for self-study prior to face-to-face (F2F) sessions. Six instructional videos, each dedicated to a specific procedure, are accessible for preview and repeated viewing as needed. Such flexibility allows the patients to revise at their own preferred time and pace.
  Participants will be asked to take note of any issues or difficulties they encounter while watching the video.
  A CAPD education booklet will be prepared and distributed to the patients at the beginning of the F2F training session.
  Take-home exercises will allow participants to revise the materials covered in the videos and consolidate their learning.
  Arms: Audio-visual assisted Flipped Classroom pre-dialysis training

SUMMARY:
The goal of this single-blinded randomized controlled trial is to evaluate the effectiveness of an educational intervention for patient self-management and successful renal replacement therapy in Chronic Kidney Disease (CKD) patients.

The main question it aims to answer is whether the flipped class pedagogy in delivering the pre-dialysis program to CKD patients is effective.

Participants will undergo a week-long intervention consisting of pre-class instructional videos, self-study tutorials, face-to-face sessions, and take-home exercises, and will be compared to those receiving the conventional educational course.

DETAILED DESCRIPTION:
The aim of this study is to examine the effectiveness of the flipped classroom approach in CAPD training for CKD patients who have to plan for receiving peritoneal dialysis therapy. Learning outcomes, adherence to therapy, occurrence of infections (episodes per patient-month) - exit site infection/tunnel infection, and PD-related peritonitis will be investigated. The ClinicalTrials.gov Identifier of this study will be applied.

Design and Randomisation This study is a single-blinded randomised controlled trial in a single centre. On completion of the baseline assessment and the screening procedure, eligible participants will be randomly assigned in equal number using sets of computer-generated random numbers into either the experimental group - FC training with audio-visual aids and the control group - Conventional Training (CT). The principal investigator and the nurse providing the intervention are aware of the patient group assignment. Assessment of the baseline and endpoints of the patient outcomes will be performed by an independent research assistant blinded to group allocation, who was not involved in the intervention. Figure 1 presented the data collection using the Consolidated Standards of Reporting Trials (CONSORT), which will be done before the commencement of the intervention (T1), immediately post-intervention (T2) and one month (T3) and three months (T4) after the completion of programme.

Participants and Study setting Patients attending the outpatient renal clinic of a Kwong Wah Hospital in Hong Kong will be approached. Stage 5 CKD patients who are planned to receive dialysis therapy will be invited to join the study. Comorbidity will not be considered in client selection since research suggested that it only explains a modest part of the variance of patient outcome in a multicenter study on CKD patients (Steenkamp, Rao, & Fraser, 2016). Eligibility for the study will be determined by the initial screening on the condition of the CKD.

ELIGIBILITY:
Inclusion Criteria:

The candidates should meet the below criteria will be recruited.

1. age ≥ 18 years
2. clinically diagnosed to have CKD Stage 5 (estimated creatinine clearance - 15 mL/min/1.73 m2)
3. Tenkoff insertion was performed and CAPD training will be offered in 4 weeks
4. able to perform self-care CAPD or family-assisted CAPD
5. willing to participate in audio-visual assisted and face-to-face activities
6. alert and oriented, able to sustain for approximately one hour of attention and interaction
7. communicable in Cantonese, able to read and write Chinese
8. could be reached by phone and able to use electronic devices, e.g. smart phone, tablet, notebook or computers to access online audio-visual materials

Exclusion Criteria:

Patients having one or above of the below conditions will be excluded from the study.

1. patients who have been receiving dialysis therapy
2. patients who are unable to communicate in Cantonese
3. patient who has hearing deficit
4. patient who are disoriented, delirious or cognitively impaired
5. patients who are clinically depressed diagnosed by medical doctors
6. patients who do not have access to online material using electronic devices
7. patients who are incompetent in giving written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Peritoneal Dialysis Psychomotor Skill Competency Checklist | Baseline assessment will be conducted prior to the intervention (T1), immediately post-intervention (T2) and one month (T3) and three months (T4) after the completion of programme.
  Patients' performance will be evaluated to see whether these are safe based on the competency checklist on peritoneal dialysis fluid exchange skills and exit site management, and the Multiple choice questions (MCQs) will be used to test the relevant knowledge.
  This assessment tool is validated by the expert panel of five members including one nephrologist, two renal nurse clinicians, and two academic staff.

SECONDARY OUTCOMES:
Student Satisfaction and Self-confidence in Learning (SSSCL) Inventory | Immediately post pre-dialysis training
  Satisfaction of the pre-dialysis programme will be measured by the Student Satisfaction and Self-Confidence in Learning (SSSCL) inventory (National League for Nursing, 2015, Chan, Fong, Tang, Gay, & Hui, 2015) to determine the satisfaction of the teaching method and self-confidence in mastering the content and skill (Cronbach's alpha from 0.87 to 0.94).
  The two subscales student satisfaction (5-items) and self-confidence (8 items) will be rated on a 5-point Likert scale scoring from strongly disagree (1) to strongly agree (5). The higher the sum scores indicate better satisfaction and self-confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Kitty Chan, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Hung Hom, Hong Kong Island, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
future multi-sites studies may be implemented, and once this is completed, and paper published, we are happy to share the IPD.
Supporting Information: Study Protocol, CSR
Time Frame: When the project is completed and publication available
Access Criteria: access by sending email to the corresponding author

REFERENCES:
- [Background] National League for Nursing. A vision for teaching with simulation: a living document from the National League for Nursing NLN Board of Governors. 2015. Retrieved from https://www.nln.org/docs/default-source/uploadedfiles/about/nln-vision-series-position-statements/vision-statement-a-vision-for-teaching-with-simulation.pdf?sfvrsn=e847da0d_0
- [Background] Chan JCK, Fong DYT, Tang JJ, Gay KP, & Hui J. The Chinese Student Satisfaction and Self-Confidence Scale Is reliable and valid. Clinical Simulation in Nursing. 2015; 11(5), 278-283. https://doi.org/10.1016/j.ecns.2015.03.003